CLINICAL TRIAL: NCT05702684
Title: Coproducing Personalised Care in a Digital Age: Using the Adversity, Restoration and Compatibility (ARC) Framework to Inform the Co-design of a Digital Care Planning Tool for People With Colorectal Cancer.
Brief Title: Personalised Cancer Care and Support: Identifying What Good Looks Like
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 312083
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People living with colorectal cancer: Patients (who are living with colorectal cancer) who have agreed to complete the eHNA intervention (within 31 days of diagnosis) and care planning consultation and clinicians who work in cancer services and provide the eHNA intervention to patients who are living with colorectal cancer
  Interventions: Other: electronic Holistic Needs Assessment (eHNA)
- People living with treatable-but-not-curable cancer: Patients who have received the ARC Holistic Needs Assessment (HNA) intervention from the ARC clinic and clinicians responsible for developing/delivering the ARC HNA intervention.
  Interventions: Other: electronic Holistic Needs Assessment (eHNA)

INTERVENTIONS:
Other: electronic Holistic Needs Assessment (eHNA) — eHNA to be completed within 31 days of diagnosis (standard care). ARC clinic previously offered 6-24 months post-diagnosis.
  Other Names: ARC clinic

SUMMARY:
The overarching aim is to study the coproduction of personalised care in a digital age by seeking to improve the experience of care and personalised care and support planning for people who live with and beyond colorectal cancer. This study will assess digital health contributions to personalised care and explore how to improve the quality of collaborative digital care planning in cancer services. The electronic holistic needs assessment (eHNA) developed by Macmillan Cancer Support (macmillan.org.uk/healthcare-professionals/innovation-in-cancer-care/holistic-needs-assessment/sign-up-to-ehna) will be used as a case study to help advance this aspect of healthcare improvement studies.

The primary objective is to gain a better understanding of how personalised care and support planning in the form of the eHNA and consultation works (or not) from the perspectives of people who are living with and beyond colorectal cancer, and clinicians.

The secondary objectives are to:

i. identify what good practice looks like for digital personalised care and support planning in a specific tumour group (colorectal) and at a point in the cancer pathway (within 31 days of diagnosis)

ii. explore if the ARC framework can be used to inform personalised cancer care and support planning

The research will review current practice and focus on identifying what good looks like for digital cancer care planning. It will go on to explore how what we know about LWBC can be used to inform the co-design of digital care planning that better supports personalised long-term cancer care. From the outset, this early work will help to inform future issues around generalisability and scaling-up.

DETAILED DESCRIPTION:
The study will use two forms of data collection: 1) Video-Reflexive Ethnography (VRE) and 2) individual interviews with patient/clinician dyads from the ARC clinic.

1. Video-reflexive ethnography Video-reflexive ethnography (VRE) is a collaborative participatory methodology used by researchers and participants, such as patients and clinicians, to understand, reflect, and improve patient experience and clinicians' work practices. Participants and researchers work together to engage with and co-construct the research, that involves three sequential phases: i) field observations of practice, ii) video recording of in-situ practice, and iii) discussing edited footage with participants in video-reflexive sessions. The film is a vital component of the process, and the critical appraisal gives participant involvement in identifying/determining the focus based on the appraisal of the real time or in-situ practice.

   i) Field observations of practice Observations of practice will be undertaken at the outset in order to capture everyday patient and staff practice and to map existing eHNA/personalised care and support planning processes and interactions (i.e., delivery and content).

   ii) Video recording of in-situ practice The research will focus on observing/filming the two components of the eHNA process by following (the same) patient-staff dyads (n=up to 15 in total across all sites) from eHNA tool to care plan. The sample size is appropriate, in terms being able to answer the research question and the methodological orientation of VRE and EBCD and the current debates on saturation.

   Component 1: Observing (in-person or virtual) patients as they interact with the eHNA

   The eHNA tool is a patient-held self-assessment, so if the patient chooses to complete the eHNA at home, the researcher will offer to host the session in-person or virtually (i.e., using zoom or MS Teams, according to their preference). Virtual observations describe a form of data collection when the researcher can witness an event that is happening online and videoconferencing (i.e., zoom) has been rated as an acceptable form of online qualitative data collection. Think aloud and question-asking techniques will be used as patients interact with the eHNA to gather user reasoning and feedback on experience as the intervention is happening. The question-asking method goes one step further than the think-aloud method, in a way that the researcher asks questions about the product being tested (eHNA tool). These methods have been successfully used in previous studies that evaluate prototypes of digital health systems. The participants do not have to tell the researcher anything about their health concerns or their medical care if they do not want to.

   Component 2: Observing (in-person or virtual) the care planning consultation with patients and clinicians

   With participant consent, the researcher will observe the care planning consultation with the (same) patient and their clinician as they review the eHNA data, conduct the care planning consultation, and complete a care plan. The observation will be video and audio-recorded to capture the interaction and to provide an opportunity to re-review the complexities of healthcare communication. The researcher's aim is to be unobtrusive, but to learn about healthcare interactions and the practices and tasks that each person is (or is not) involved in as part of personalised care and support planning. The consultation forms a component of the eHNA process and is offered to all patients as standard care. The consultation meeting is usually organised by the clinician and conducted in a private 1:1 space. If the clinical interaction is conducted virtually (i.e., a zoom consultation), the researcher will join the meeting virtually. If the consultation is conducted by telephone, the researcher will either join the meeting from the NHS Trust site and the consultation will take place by speakerphone in a private room.

   Alternatively, the researcher will join the meeting with the patient, according to patient preference. The researcher will not speak during observations unless participants have questions about the study.

   iii) Video-reflexive sessions with a) patients, b) clinicians, and c) teams

   The research team/chief investigator will edit clips from the two videos into a short 5-10 minute film. Patients will be asked to attend a video-recorded reflexive session to review the video footage and reflect on their eHNA and care planning experience. They will be asked to reflect on what has gone well and what could be improved. This session will take place at home or in a private room at the NHS Trust site where the patient receives their care. If the patient chooses to have the session at home, the researcher will offer to host the session in-person or virtually (i.e., using zoom or MS Teams, according to their preference).

   Clips from the three videos (i) patient as they interact with the eHNA tool, ii) care planning consultation, iii) patient reflexive session will then be edited into one short film by the research team. The edited film will be shared with the paired clinician to allow them to also reflect on what went well and on what could be improved, and to learn from the experience in a clinician reflexive session. All video clips intended for the team reflexivity sessions will be shared with the patient/clinician to ensure they are happy for the chosen clips to be shown. In this way, the patient/clinician can also be involved in identifying topics for analysis and selecting the clips to be shown to teams. The edited video provides a concentrated focus to generate conversation and to gain in-depth insight into experiences of practice. In this way, VRE works as a catalyst for healthcare practice change. The researcher is also actively involved in the process as a co-creator, that is, leading the editing of video clips and facilitating the reflexive sessions. The staff and team reflexive sessions will last approximately 60-90 minutes and will take place either face-to-face at the NHS Trust site where the clinician/team works or online, depending on preference. The session will be led by a researcher and will be audio-recorded in order to capture all experiences, views, and ideas accurately. Before all reflexivity sessions, the edited clips are reviewed by those featured in footage and the specific time and place for the reflexivity sessions are decided in negotiation with the participants. The focus of the clinician/team reflexive sessions is for staff to learn from each other (with the help of VRE), to identify strengths of practice as well as opportunities for improvement.
2. Individual interviews with patient/clinician dyads from the ARC clinic (in-person or virtual depending on participant preference and/or covid-19 regulations)

Interview data meets the research aim by capturing perspectives, attitudes, and values in relation to personalised care and support planning. Semi-structured individual interviews will explore experiences of attending/working in the ARC clinic, perspectives on the value of the ARC clinic intervention, areas for improvement, and will allow for overall reflection of being involved in the ARC clinic project/their experience of care. As this is an investigative study, individuals will be encouraged to tell their own story and to share their views, attitudes, experiences, and perceptions in an open way. Patients (n=5) and clinicians (n=3) will be interviewed separately and not together as a pair.

ELIGIBILITY:
Inclusion Criteria:

Patients

1. Patients (who are living with and beyond colorectal cancer) who have agreed to complete the eHNA intervention within 31 days of diagnosis OR patients who received the ARC clinic HNA intervention.
2. Over 18 years of age
3. Speak a conversational level of English Patients will be sampled purposively to ensure a range of experiences. Patients will be sampled on ethnicity, gender, age, time since diagnosis, socio-economic status, and digital maturity, so that findings can also be used to explore and address cancer inequalities.

Paired clinicians

1. Clinicians (e.g., CNS, AHP, cancer support worker) who work in cancer services and provide the eHNA/ARC intervention to (the recruited) patients who are living with colorectal cancer.
2. Over the age of 18
3. Speak a conversational level of English.

Team members

1. Clinicians (e.g., CNS, AHP, cancer support worker) who work in the colorectal cancer team or who work in close liaison with the colorectal cancer team and are responsible for providing the eHNA and care planning consultation.
2. Over the age of 18
3. Speak a conversational level of English.

Exclusion Criteria:

Patients

1. Patients (who are living with and beyond cancer) who are receiving treatment but who have not agreed to complete an eHNA /patients who did not attend the ARC clinic.
2. Under 18 years of age
3. Do not speak a conversational level of English
4. Patients who lack capacity to consent

Patients that are approached to take part in the study but who do not want to participate will automatically be excluded from the project. Insufficient ability to understand/speak English is an exclusion criterion for this study because the research uses audio recordings of verbal conversation and relies on understanding of written study materials in order to ensure informed consent. Participants with a low level of literacy (but with adequate conversational level of English) can be supported by having the researcher read out the participant information sheet and consent form, and to check for understanding.

Paired Clinicians 1. Clinicians who do not provide the eHNA intervention /ARC intervention to patients who are living with and beyond cancer.

Team members

1. Clinicians (e.g., CNS, AHP, cancer support worker) who do not work in the colorectal cancer team or in close liaison with the colorectal cancer team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will focus on colorectal (including metastatic disease but not end of life) cancer. This group of patients have immediate needs (i.e., body image, disruption in life), and require ongoing treatment (up to 15 years of treatment options). This tumour group also has a fairly equal age and gender distribution and is underrepresented in research (Sun et al., 2021). Changes to colorectal cancer care delivery during the COVID-19 pandemic have also shown to increase healthcare inequalities (Ip et al., 2022). The study will focus on the eHNA process at diagnosis (within 31 days of diagnosis) because this is already a focus for services in terms of meeting NHS England key performance indicators.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Patient experience | Through study completion up to 12 months
  Improved experience of care as measured through video-reflexive ethnography processes

CONTACTS AND LOCATIONS:
Overall Officials: Clair Le Boutillier, Principal Investigator — King's College London
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study is compliant with the requirements of General Data Protection Regulation (2016/679) and the Data Protection Act (2018). All investigators and study site staff will comply with the requirements of the General Data Protection Regulation (2016/679) with regards to the collection, storage, processing, and disclosure of personal information, and will uphold the Act's core principles. The sponsors for this study will be King's College London (KCL) and Guys and St Thomas' NHS Foundation Trust (GSTT). KCL and GSTT are joint data controllers.

REFERENCES:
- [Background] Carroll K, Mesman J. Multiple Researcher Roles in Video-Reflexive Ethnography. Qual Health Res. 2018 Jun;28(7):1145-1156. doi: 10.1177/1049732318759490. Epub 2018 Feb 24. PMID 29478407
- [Background] Wyer M, Jackson D, Iedema R, Hor SY, Gilbert GL, Jorm C, Hooker C, O'Sullivan MV, Carroll K. Involving patients in understanding hospital infection control using visual methods. J Clin Nurs. 2015 Jun;24(11-12):1718-29. doi: 10.1111/jocn.12779. Epub 2015 Feb 7. PMID 25662176
- [Background] Iedema R. Research paradigm that tackles the complexity of in situ care: video reflexivity. BMJ Qual Saf. 2019 Feb;28(2):89-90. doi: 10.1136/bmjqs-2018-008778. Epub 2018 Oct 11. No abstract available. PMID 30309911
- [Background] Varpio L, Ajjawi R, Monrouxe LV, O'Brien BC, Rees CE. Shedding the cobra effect: problematising thematic emergence, triangulation, saturation and member checking. Med Educ. 2017 Jan;51(1):40-50. doi: 10.1111/medu.13124. PMID 27981658
- [Background] Iedema RA, Angell B. What are patients' care experience priorities? BMJ Qual Saf. 2015 Jun;24(6):356-9. doi: 10.1136/bmjqs-2015-004298. Epub 2015 May 13. No abstract available. PMID 25972222